CLINICAL TRIAL: NCT00647946
Title: A Phase II, Open-Label, Multicentre, Randomised, Comparator Study of Substitution With Tenofovir or Abacavir in HIV-1 Infected Individuals, With a Viral Load < 50 Copies/mL, Receiving a Thymidine Analogue (Zidovudine or Stavudine) as Part of Their Highly Active Antiretroviral Therapy (HAART)
Brief Title: Study to Evaluate Changes in Limb Fat When Switching From a Thymidine Analogue
Acronym: RAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Geoff Cotton, Medical Monitor, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-UK-104-1008
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Lipodystrophy
Keywords: lipodystrophy
MeSH Terms: conditions — Lipodystrophy | interventions — Tenofovir; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Stop zidovudine (ZDV) or stavudine (d4T) and start tenofovir DF 300mg once daily along with the other antiviral drugs that are used as part of their HAART regimen
  Interventions: Drug: tenofovir DF
- B (Active Comparator): Stop zidovudine (ZDV) or stavudine (d4T) and start abacavir 300mg twice daily along with the other antiviral drugs that are used as part of their HAART regimen
  Interventions: Drug: abacavir 300mg twice daily

INTERVENTIONS:
Drug: tenofovir DF — tenofovir DF 300mg once daily along with the other antiviral drugs
  Arms: A
Drug: abacavir 300mg twice daily — abacavir 300mg twice daily along with the other antiviral drugs
  Arms: B

SUMMARY:
A previous study substituting zidovudine or stavudine to abacavir in patients with severe or moderate lipoatrophy has shown an increase in limb fat by DEXA. This study was conducted over a 24-week period and although improved outcomes were documented by objective measures, DEXA scans, subjective observation did not correspond. Longer-term follow up of these patients is required.

This 48 week study is designed to compare the substitution of the thymidine analogues zidovudine (ZDV) or stavudine (D4T) with either tenofovir DF or abacavir, in patients treated with highly active antiretroviral therapy (HAART), and show improved outcomes on total limb fat mass, improved body shape by dual energy x-ray absorptiometry (DEXA) and computed tomography (CT) scans and improved cholesterol and triglycerides.

DETAILED DESCRIPTION:
This is a phase II, open-label, multicentre, randomised, two-arm study of 48 weeks duration. One hundred HIV infected individuals who have documented lipodystrophy at > 1 body/facial site and currently receiving zidovudine (ZDV) or stavudine (d4T) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are male or female > 18 years of age
* Subjects who are HIV-1 infected as documented by a licensed HIV-1 antibody ELISA
* Female subjects of childbearing potential must have a negative serum pregnancy test (beta-HCG) within 28 days of trial day 1. Women of childbearing potential must agree to use a barrier method of contraception
* Female subjects must not be pregnant or lactating
* Subjects who in the opinion of the investigator have the ability to understand and provided written informed consent to participate in the trial
* Subjects who in the opinion of the investigator have clinical lipoatrophy at > 1 body/facial site
* Subjects currently receiving nucleoside analogue regimen including stavudine (d4T) or zidovudine (ZDV)
* Subjects who are stable on current therapy for >16 weeks
* Subjects with no prior exposure to tenofovir, abacavir, or adefovir
* Subjects with no known K65R, 69S mutations or 3 or more thymidine analogue mutations
* Subjects with documented viral load <50 copies/ml on 2 consecutive occasions including most recent clinic attendance

Exclusion Criteria:

* Subjects who in the investigator's opinion are unlikely to complete the 48 week trial period
* Currently active opportunistic disease or documented wasting syndrome
* Currently receiving chemotherapy for malignancy
* Subjects who in the opinion of the investigator are unlikely to retain viral response after switching based on treatment or transmission history
* Currently receiving an insulin sensitising agent (glitazone or metformin)
* Anabolic steroids in the last 16 weeks other than testosterone at replacement doses (<250mg/2 weekly)
* Growth hormone use in the last 16 weeks
* Statin therapy (HMG CoA reductase inhibitor) commenced in the last 16 weeks (patients stable on statins my be included)
* Current alcohol or illicit drug use which, in the opinion of the investigator, may interfere with the subjects' ability to comply with the dosing schedule and protocol evaluations
* Receiving concurrent medications that - in the opinion of the investigator and according to drug product labelling - will result in clinically significant interactions with tenofovir or abacavir
* Pregnant or breast feeding
* Previously received more than 3 months zidovudine monotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-02; Primary Completion 2004-10 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change in total limb fat mass by DEXA scan | 24 and 48 weeks

SECONDARY OUTCOMES:
Change in VAT by single slice L4 abdominal CT scan | 24 and 48 weeks
Change in viral load measurements and CD4 cell count | 24 and 48 Weeks
Change in fasting cholesterol and triglycerides | 24 and 48 Weeks
Change in blood insulin and fasting glucose | 24 and 48 Weeks
Change in blood lactate and anion gap | 24 and 48 Weeks
Change in bone mineral density by DEXA scan | 24 and 48 Weeks
Incidence of adverse events | Upto 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Cotton, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Abingdon, Cambridge, United Kingdom

REFERENCES:
- See also: Study results — http://www.gileadclinicaltrials.com/